CLINICAL TRIAL: NCT02566590
Title: Preventing the Loss of Muscle and Function in Hospitalized Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Micah Drummond, Ph.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 72083
Record Dates: First submitted 2015-09-23; First posted 2015-10-02 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2018-10

CONDITIONS: Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy | interventions — Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Experimental): Participants will complete bed rest but will receive a non-protein placebo supplement
  Interventions: Dietary Supplement: non-protein placebo supplement
- NMES + PRO (Experimental): Participants will receive daily treatment with neuromuscular electrical stimulation (NMES) and daily supplements of a protein drink.
  Interventions: Device: NMES; Dietary Supplement: Protein

INTERVENTIONS:
Device: NMES — device is used to stimulate muscle contraction in the legs of the patient. The intervention will be used 3 times a day during bed rest.
  Arms: NMES + PRO
Dietary Supplement: Protein — supplement will used to enhance muscle anabolism. The intervention will be provided 3 times a day during bed rest.
  Arms: NMES + PRO
Dietary Supplement: non-protein placebo supplement — supplement will be used as a placebo to control participants. The supplement will be provided 3x a day during bed rest.
  Arms: Control

SUMMARY:
One third of independent older adults over the age of 65y will be hospitalized for an acute medical illness, injury, or operative procedure. Unfortunately, 50% of these older adults will experience functional decline during their hospital stay from the amount of time they are physically inactive and in bed. Following discharge, the functional deficits can persist for months and in many instances never return to pre-hospitalization levels thus compounding morbidity, health care costs and dying. A classic consequence of short-term bed rest in older adults is the significant loss in skeletal muscle mass which underlies the accelerated leg strength deficits. The investigator has shown that an important mechanism of skeletal muscle loss is the inability of nutrients to stimulate a normal muscle protein synthesis response; a process highly regulated by the mammalian target of rapamycin signaling pathway (mTOR) and amino acid transporters. Day to day maintenance of force generating muscle tissue is dictated by anabolic stimulation from muscle contraction and essential amino acid ingestion. Therefore, anabolic interventions such as neuromuscular electrical stimulation (NMES) and high quality protein supplementation that contains a high proportion of essential amino acids (whey protein) may be promising approach to maintain leg muscle mass and strength in hospitalized older adults and prevent the long term consequences of repeated periods of short-term physical inactivity. The purpose of this study is to test in older adults if the combination of NMES and protein supplementation is capable of preserving muscle mass and strength and maintaining muscle nutrient anabolic sensitivity during bed rest. The investigators current hypotheses are that daily NMES and protein supplementation during 5-days of bed rest in older adults will: 1) preserve lower extremity muscle mass and strength and 2) maintain muscle nutrient anabolic sensitivity as measured by mTOR signaling and amino acid transporter expression. The long term goal is to utilize this inpatient preventative therapeutic approach in a clinical setting in which muscle mass and strength deficits are profound (e.g., intensive care patients).

DETAILED DESCRIPTION:
A majority of older adults experience repeated periods of physical inactivity during acute illnesses, injuries or after an operative procedure. Following discharge from the hospital, daily activities are adversely impacted. Infirmity follows repeated periods of inactivity (termed "catabolic hits") that can occur over an older adults' lifespan and lead to a downward spiral of potentially irrecoverable deficits in physical function resulting in increased health care costs, loss of independence, and premature death. The hallmark sign of short-term physical inactivity in older adults is the rapid deterioration of skeletal muscle mass and strength. Understandably, little attention is placed on physical function during these requisite periods of inactivity as the medical management and/or postoperative recuperation is the focus. However, the muscle deficits that follow as a result of acute hospitalization can have profound long-term consequences.

Muscle contraction and essential amino acids are powerful independent anabolic stimuli and fundamental to maintain skeletal muscle mass and strength. The primary mechanism of disuse atrophy during short-term bed rest in older adults is the reduced acute nutrient stimulation of muscle protein synthesis regulated by the mammalian target of rapamycin (mTOR) signaling pathway and amino acid transporter expression (i.e., LAT1). Intervening with essential amino acid supplements can maintain some muscle function in older adults during bed rest, but it does not preserve muscle mass. Neuromuscular electrical stimulation (NMES) as a muscle intervention is also feasible, but alone is not a panacea. NMES has recently been shown to acutely stimulate protein synthesis in ambulatory older adults with diabetes and attenuate some loss in muscle mass in critically ill patients. The investigator suggests that, together, daily NMES, and a high quality protein source of EAAs (PRO), can be a potent two-pronged approach to preserve the loss of muscle and strength in older adults confined to short-term bed rest. The goal is to test if the combination of NMES and PRO will maintain muscle mass, strength, nutrient-induced mTOR signaling and amino acid transporter expression in older adults during bed rest. The central hypothesis for this project which will support this next step is that a daily combination of NMES and PRO in older adults experiencing bed rest will preserve: 1) leg muscle mass and knee extensor strength and 2) muscle anabolic sensitivity in response to acute nutrient ingestion, as measured by mTOR signaling and LAT1 expression.

ELIGIBILITY:
Inclusion Criteria:

Age between 60-85 yrs Ability to sign informed consent Montreal cognitive assessment (MOCA) exam score ≥26 Free-living, prior to admission

Exclusion Criteria:

1. Cardiac abnormalities considered exclusionary by the study physician (e.g., CHF, CAD, right-to-left shunt)
2. Uncontrolled endocrine or metabolic disease (e.g., hypo/hyperthyroidism, diabetes)
3. GFR <65 mL/min/1.73m2 or evidence of kidney disease or failure
4. Vascular disease or risk factors of peripheral atherosclerosis. (e.g., uncontrolled hypertension, obesity, diabetes, hypercholesterolemia > 250 mg/dl, claudication or evidence of venous or arterial insufficiency upon palpitation of femoral, popliteal and pedal arteries)
5. Risk of DVT including family history of thrombophilia, DVT, pulmonary emboli, myeloproliferative diseases including polycythemia (Hb>18 g/dL) or thrombocytosis (platelets>400x103/mL), and connective tissue diseases (positive lupus anticoagulant), hyperhomocysteinemia, deficiencies of factor V Leiden, proteins S and C, and antithrombin III
6. Use of anticoagulant therapy (e.g., Coumadin, heparin)
7. Elevated systolic pressure >150 or a diastolic blood pressure > 100
8. Implanted electronic devices (e.g., pacemakers, electronic infusion pumps, stimulators)
9. Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
10. Currently on a weight-loss diet or body mass index > 30 kg/m2
11. Inability to abstain from smoking for duration of study
12. A history of > 20 pack per year smoking
13. HIV or hepatitis B or C*
14. Recent anabolic or corticosteroids use (within 3 months)
15. Subjects with hemoglobin or hematocrit lower than accepted lab values
16. Agitation/aggression disorder (by psychiatric history and exam)
17. History of stroke with motor disability
18. A recent history (<12 months) of GI bleed
19. Depression [>5 on the 15 items Geriatric Depression Scale (GDS)]
20. Alcohol or drug abuse
21. Exercise training (>1 session of moderate to high intensity aerobic or resistance exercise/week)
22. Liver disease (AST/ALT 2 times above the normal limit, hyperbilirubinemia)
23. Respiratory disease (acute upper respiratory infection, history of chronic lung disease with resting oxygen saturation <97% on room air)
24. Any other condition or event considered exclusionary by the PI and faculty physician

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micah Drummond, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | NMES + PRO
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | NMES + PRO | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6.7) | 69 (5.4) | 69 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Percent Change in Bilateral Thigh Lean Mass Density (Grams) as Measured by DEXA Scan Will be Compared Between Baseline and After 5-days of Bed Rest
Description: Thigh lean mass (grams) will be measured by DEXA scan at baseline and after 5-days of bed rest. The change in thigh lean mass will be calculated between these two time points. This outcome will be measured for the Control and the NMES + PRO groups.
Time Frame: Baseline and after 5-days of Bed rest
Measure: Mean (Standard Error); unit: Percent Change
Groups:
- Control: Participants will complete bed rest but will receive a non-protein placebo supplement
  non-protein placebo supplement: supplement will be used as a placebo for control participants. The supplement will be provided 3x a day during bed rest.
- NMES + PRO: Participants will receive daily treatment with neuromuscular electrical stimulation (NMES) and daily supplements of a protein drink.
  NMES: device is used to stimulate muscle contraction in the legs of the patient. The intervention will be used 3 times a day during each day of bed rest.
  Protein (PRO): supplement will used to enhance muscle anabolism. The intervention will be provided 3 times a day during each day of bed rest.
Arm/Group | Control | NMES + PRO
Number analyzed (Participants) | 10 | 10
Percent Change | -3.845 (0.883) | -0.249 (1.189)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Control | NMES + PRO
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No